CLINICAL TRIAL: NCT06122688
Title: By Youth, For Youth: Digital Supported Peer Navigation for Addressing Child Mental Health Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Riverside (Other)
Collaborators: University of California, San Francisco (Other); University of California, Los Angeles (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: U01MH131827 (NIH)
Record Dates: First submitted 2023-10-31; First posted 2023-11-08 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Depression; Mental Health Issue
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: In each county, 10 sites will participate (10 high schools in Los Angeles and 10 Primary Care Clinics in Riverside), with sites randomized to cross over from control to intervention status in a step wedged design each Fall following the beginning of the school year. Three months is allowed for training and setup at each site prior to intervention delivery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care as usual (No Intervention): All individuals within each site regardless of type of site or step period will begin with a control period of care as usual
  Youth and parents within each site will have access to navigators who will share information about mental health and social services supports as well as referrals.
  The duration of the control period (1, 2, or 3 years; collected via medical and/or other administrative records) will depend on the step period of the individual's site.
- Implementation (Experimental): In this stepped wedge design, following a period of care as usual as a control, sites will then cross over to the experimental arm, during which, all youth and their caregivers at the enrolled site are encouraged to download and use the wellness app for the duration of the implementation period. Navigators promote and support use of the app.
  Interventions: Behavioral: Navigator Plus App Intervention

INTERVENTIONS:
Behavioral: Navigator Plus App Intervention — Navigators will provide their usual care services and also be encouraged to use the Connected for Wellness (CFW) app during their usual activities with youth and caregivers at their site. The duration of this period (2, 3, or 4 years) will depend on the step period of the individual's site. All youth at the school or clinic site can use the CFW app on their own and through the app receive prevention strategies, psycho-education that destigmatizes mental health, encourages referrals to local resources as needed, and increases motivation to access care if needed.
  Arms: Implementation

SUMMARY:
Despite significant progress in research, practice, and policy over the past few decades, many children and youth continue to experience poor mental health outcomes. With their unrivaled ability to reach youth, school-based services and primary care are ideal hubs to provide mental health, healthcare, social services, and prevention to youth and families who otherwise face barriers to care. Using Participatory Design and Community Partnered Participatory Research (CPPR) for app development, mobile technology is designed to optimize access to wellness resources. The proposed intervention is a model of care using technology and navigators for connecting youth ages 13-22 to mental health care and supports. The app is co-created with the community and supported by culturally responsive individuals called family and youth navigators, in schools and primary care clinics. Outcomes are measured using the cascade of care model.

DETAILED DESCRIPTION:
Using Participatory Design and Community Partnered Participatory Research (CPPR), UCLA and UCR psychiatry research centers with Los Angeles Trust for Children's Health aim to: (1) Fully co-design (with youth, caregivers, clinicians and other stakeholders) an innovative mental health digital tool, called Connected for Wellness, to implement algorithmically supported mental health + social determinants, resiliency app based tools and navigation activities AND help support the clinical workforce within schools and primary care clinics (PCCs); (2) Study the implementation of mental health navigation models (family and youth navigation) plus the Connected for Wellness app, and their effectiveness for improving connecting and matching youth to the right level of care and supports. We will accomplish these aims through three strategies: (1) Use community participatory informatics to co-design a mental health digital tool called Connected for Wellness, to support mental health navigation, linking youth to a range of mental health services, evidence-based prevention resources referred via the app, and other school, clinic, community, and social supports; (2) Integrate mental health self-assessments and artificial intelligence (AI) in Connected for Wellness to individualize app resources, optimize engagement and recommendations for addressing mental health and social needs; (3) Using a stepped wedge design, test the implementation of the app supported by mental health navigation models (peer navigators, family navigators) for improving connections and access to prevention resources, mental health services and social supports, for youth and families. This project will be initiated with youth 13-22 years old and their family and community members across 10 Los Angeles County Schools and 10 Riverside County/University of California Riverside primary care clinics. A successful outcome of the project is a CPPR developed app-based intervention implementable in school-based and primary care services for access to wellness resources and improving mental health services access along the cascade of care. Outcomes are measured using the cascade of care model with the following key stages: (1) need identification, (2) referral to care/ linkage to resources, and (3) care initiation.

ELIGIBILITY:
Inclusion Criteria:

* Youth 13-22 enrolled in high school or participating primary care clinics, and their caregivers.

Exclusion Criteria:

* Those not meeting inclusion criteria

Ages: 13 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8360 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of youth referred to mental health services who initiate care. | 1 year
  Referral to and initiation of mental health services data will be obtained from electronic medical records.

SECONDARY OUTCOMES:
Proportion of youth completing a mental health screening who are referred to care. | 1 year
  Mental health screening and referral to mental health services data will be obtained from electronic medical records.

OTHER OUTCOMES:
Proportion of youth in school/clinic completing a mental health screening. | 1 year
  Mental health screening data will be obtained from electronic medical records.
Proportion of youth initiating mental health services who have 3 or more visits. | 1 year
  Mental health initiation and visit data will be obtained from electronic medical records.

REFERENCES:
- [Background] Cook BL, Trinh NH, Li Z, Hou SS, Progovac AM. Trends in Racial-Ethnic Disparities in Access to Mental Health Care, 2004-2012. Psychiatr Serv. 2017 Jan 1;68(1):9-16. doi: 10.1176/appi.ps.201500453. Epub 2016 Aug 1. PMID 27476805
- [Background] Marrast L, Himmelstein DU, Woolhandler S. Racial and Ethnic Disparities in Mental Health Care for Children and Young Adults: A National Study. Int J Health Serv. 2016 Oct;46(4):810-24. doi: 10.1177/0020731416662736. Epub 2016 Aug 12. PMID 27520100
- [Background] Kataoka SH, Vona P, Acuna A, Jaycox L, Escudero P, Rojas C, Ramirez E, Langley A, Stein BD. Applying a Trauma Informed School Systems Approach: Examples from School Community-Academic Partnerships. Ethn Dis. 2018 Sep 6;28(Suppl 2):417-426. doi: 10.18865/ed.28.S2.417. eCollection 2018. PMID 30202195
- [Background] Arevian AC, Jones F, Moore EM, Goodsmith N, Aguilar-Gaxiola S, Ewing T, Siddiq H, Lester P, Cheung E, Ijadi-Maghsoodi R, Gabrielian S, Sugarman OK, Bonds C, Benitez C, Innes-Gomberg D, Springgate B, Haywood C, Meyers D, Sherin JE, Wells K. Mental Health Community and Health System Issues in COVID-19: Lessons from Academic, Community, Provider and Policy Stakeholders. Ethn Dis. 2020 Sep 24;30(4):695-700. doi: 10.18865/ed.30.4.695. eCollection 2020 Fall. PMID 32989370
- [Background] Balcombe L, De Leo D. Digital Mental Health Challenges and the Horizon Ahead for Solutions. JMIR Ment Health. 2021 Mar 29;8(3):e26811. doi: 10.2196/26811. PMID 33779570
- [Background] Ellis DM, Draheim AA, Anderson PL. Culturally adapted digital mental health interventions for ethnic/racial minorities: A systematic review and meta-analysis. J Consult Clin Psychol. 2022 Oct;90(10):717-733. doi: 10.1037/ccp0000759. Epub 2022 Oct 13. PMID 36227330
- [Background] Fortuna LR, Tolou-Shams M, Robles-Ramamurthy B, Porche MV. Inequity and the disproportionate impact of COVID-19 on communities of color in the United States: The need for a trauma-informed social justice response. Psychol Trauma. 2020 Jul;12(5):443-445. doi: 10.1037/tra0000889. Epub 2020 Jun 1. PMID 32478545
- [Background] Lyon AR, Koerner K. User-Centered Design for Psychosocial Intervention Development and Implementation. Clin Psychol (New York). 2016 Jun;23(2):180-200. doi: 10.1111/cpsp.12154. Epub 2016 Jun 17. PMID 29456295
- [Background] Park SY, Nicksic Sigmon C, Boeldt D. A Framework for the Implementation of Digital Mental Health Interventions: The Importance of Feasibility and Acceptability Research. Cureus. 2022 Sep 19;14(9):e29329. doi: 10.7759/cureus.29329. eCollection 2022 Sep. PMID 36277565
- [Background] Porche MV, Folk JB, Tolou-Shams M, Fortuna LR. Researchers' Perspectives on Digital Mental Health Intervention Co-Design With Marginalized Community Stakeholder Youth and Families. Front Psychiatry. 2022 Apr 22;13:867460. doi: 10.3389/fpsyt.2022.867460. eCollection 2022. PMID 35530032
- [Derived] Fortuna LR, Porche MV, Shumway M, Ijadi-Maghsoodi R, Aralis H, Folk JB, Tolou-Shams M, Barish G, Gonzalez JC, Kataoka S. Addressing Youth Mental Health Through Schools and Primary Care Clinics Using the Connected for Wellness Mobile App: Protocol for a Stepped-Wedge Trial. JMIR Res Protoc. 2025 Aug 26;14:e73721. doi: 10.2196/73721. PMID 40857099